CLINICAL TRIAL: NCT04216303
Title: Optimal A1c Control in Post Liver or Combined Liver and Kidney Transplant Recipients Who Have Diabetes Mellitus
Status: Withdrawn | Type: Observational
Why Stopped: PI decided to stop the study
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 037.IMD.2019.D
Record Dates: First submitted 2019-09-12; First posted 2020-01-02 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Diabetes; Liver Transplant; Complications; Kidney Transplant Failure
Keywords: hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: hemoglobin A1c — The hemoglobin A1c test (A1c) screens for, helps diagnose, and monitors diabetes and prediabetes.

SUMMARY:
Major cardiovascular events are greatest in liver transplant recipients with sustained post-transplantation diabetes1. However, the optimal A1c target after transplantation has not been studied. The objective is to understand the optimal A1c target post liver and combined liver and kidney transplant. Strict A1c control will improve mortality and cardiovascular risk post liver and combined liver and kidney transplant and improve complications post liver and combined liver and kidney transplant.

DETAILED DESCRIPTION:
Major cardiovascular events are greatest in liver transplant recipients with sustained post-transplantation diabetes. However, the optimal A1c target after transplantation has not been studied. The objective is to understand the optimal A1c target post liver and combined liver and kidney transplant. Strict A1c control will improve mortality and cardiovascular risk post liver and combined liver and kidney transplant and improve complications post liver and combined liver and kidney transplant.

Strict blood sugar control in non-transplant patients with diabetes mellitus has shown unfavorable results in previous studies. However, no optimal A1c level has been studied in liver and combined liver and kidney transplant patients. Furthermore, guidelines for A1c target post-transplant are of expert opinion.

The primary objective is to assess the impact of hemoglobin A1c on all-cause mortality among patients with diabetes mellitus undergoing liver or combined liver and kidney transplantation between 2008 to 2018. The second objective is to assess the impact of hemoglobin A1c on complications post liver or combined liver and kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years old or older in the United States with diabetes undergoing or post liver and combined liver and kidney transplant from January 2008 to December 2018.

Exclusion Criteria:

* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be obtained from UNOS, which is a large, non-profit organization, database about organ transplant recipients in the United States. Data will be collected from January 2008 to December 2018, and compared outcomes (as mentioned above) between liver and combined liver and kidney transplant recipients with A1c values <6.0, 6.1 to 7.0, 7.1 to 8.0, 8.1 to 8.9, or >9.0.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-08-19 (Estimated); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Stroke or myocardial infarction | January 2008 to December 2018
cause specific mortality from infection/sepsis | January 2008 to December 2018

CONTACTS AND LOCATIONS:
Overall Officials: Mangesh Pagadala, MD, Principal Investigator — The Liver Institute Methodist Dallas Medical Center
Locations (1):
- Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided